CLINICAL TRIAL: NCT00479180
Title: Safety of Vascugel Treatment After Creation of Arteriovenous Access for Hemodialysis Use
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pervasis Therapeutics, Inc (Industry)
Responsible Party: Elizabeth Merica, Director,Clinical Affairs, Pervasis Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVS-06-003/06-004
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Hemodialysis Access
Keywords: Hemodialysis access; Arteriovenous graft; Arteriovenous fistula; End stage renal disease
MeSH Terms: conditions — Arteriovenous Fistula; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AVG1 (Experimental): Vascugel
  Interventions: Biological: Vascugel
- AVG2 (Placebo Comparator): Gelfoam
  Interventions: Biological: Placebo Comparator
- AVF3 (Experimental): Vascugel
  Interventions: Biological: Vascugel
- AVF4 (Placebo Comparator): Gelfoam
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: Vascugel — One time implant on the day of surgery
  Arms: AVF3; AVG1
Biological: Placebo Comparator — One time implant on the day of surgery
  Arms: AVF4; AVG2

SUMMARY:
Vascugel™ is safe when placed at the anastomotic site at the time of surgery during creation of an AV graft or fistula for hemodialysis access.

DETAILED DESCRIPTION:
Randomized, double-blind, parallel group, Phase I/II clinical trial of Vascugel™ treatment vs. Gelfoam® in patients undergoing creation of an arteriovenous graft or fistula for hemodialysis access.

All patients will undergo preoperative duplex ultrasound imaging and/or angiography (whatever is the standard of care at the research site) of the vein and artery to evaluate the optimal site for vascular access placement in the upper extremity.

Patients will be examined with Doppler ultrasound or standard of care immediately after surgery to verify patency of the AV graft or fistula.

During the follow-up period, each patient will undergo a physical examination and imaging of the vascular access at specified intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients (ages of 18 to 89, inclusive) who are undergoing placement of an AV graft or fistula for hemodialysis access

Exclusion Criteria:

* Patient is currently on an active transplant list for a kidney from a deceased donor OR is undergoing assessment and expects to be placed on the active transplant list within the next twenty-four weeks OR expects to receive a living donor kidney within twenty-four weeks.
* Patient is expecting another solid organ transplant or a bone marrow transplant.
* Patient has had more than one access surgery (defined as a new access, not a revision) in the target limb.
* Patient is currently on chronic, systemic immunosuppressant medication other than locally or topically applied steroids.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety of vascugel | 6 months followed by 2.5 year extension

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States